CLINICAL TRIAL: NCT00938873
Title: Understanding the Impact of Meditative Homework on Metacognitive Processes in the Context of Mindfulness Based Cognitive Therapy (MBCT)
Status: Completed | Type: Observational
Sponsor: Lahtinen, Marika (Other)
Collaborators: University of East London (Other); South London and Maudsley NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Marika Lahtinen, Dr, University of East London
Other Study IDs: 1-Lahtinen
Record Dates: First submitted 2009-07-13; First posted 2009-07-14 (Estimated); Last update posted 2012-02-29 (Estimated); Status verified 2012-02

CONDITIONS: Depression
Keywords: MBCT; identity; depression; recurrent; homework
MeSH Terms: conditions — Depression; Recurrence | interventions — Mindfulness-Based Cognitive Therapy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Mindfulness Based Cognitive Therapy: The present study will use participants who have experienced more than three episodes of depression as judged by South London and Maudsley NHS Trust. No restrictions are placed in terms of participants' use of antidepressant medication. Participants will be 18 to 65 years old and would have participated in an MBCT course run by South London and Maudsley NHS Trust.
  Interventions: Behavioral: Mindfulness Based Cognitive Therapy (MBCT)

INTERVENTIONS:
Behavioral: Mindfulness Based Cognitive Therapy (MBCT) — Mindfulness based cognitive therapy (MBCT) is a group psycho-educational treatment designed to reduce the risk of recurrent depression by integrating mindfulness based meditation practices with cognitive therapy techniques. MBCT comprises eight weekly two-hour group sessions with an additional one hour daily 6 days a week for meditative homework practice.
  Other Names: MBCT

SUMMARY:
Mindfulness based cognitive therapy (MBCT) is a group psycho-educational treatment designed to reduce the risk of recurrent depression by integrating mindfulness based meditation practices with cognitive therapy techniques. MBCT comprises eight weekly two-hour group sessions. Additionally, participants are required to commit to one hour per day of between sessions meditative homework assignments six days per week. Existing quantitative research suggest that MBCT is an effective intervention for preventing depressive relapse in patients with three or more episodes of depression (Teasdale et al.2000, Ma & Teasdale, 2004). The focus of qualitative research has been on evaluating the acceptability of MBCT for various clinical populations; participants' accounts have been positive indicating MBCT may be a potential therapeutic tool for treating older adults (Graham & Senthinathan, 2007), psychosis (Abba, Chadwick, & Stevenson, 2008), Parkinson's disease (Fitzpatrick, Simpson, & Smith, 2010) as well as acute depression (Mason & Hargreaves, 2001).

The benefits of undertaking meditative mindfulness practice in the context of MBCT have been linked to changes in metacognitive processes. Two distinct multi-level information processing frameworks dealing with how thoughts are processed from a metacognitive perspective have been proposed: The Interacting Cognitive Subsystems (ICS; Teasdale, 1999a, 1999b) and the Self Regulatory Executive Function (S-REF; Wells, 2000) theory. The ICS framework forms a rationale for meditative aspects of the MBCT programme. The S-REF model differs from the ICS theory in its conceptualisation of the object or 'being' mode of metacognitive processing.

Regular daily practice of mindfulness meditation has been regarded as among the most essential aspects of mindfulness programmes (Kabat-Zinn, 1990; Mason & Hargreaves, 2001). Existing studies, with their focus on effectiveness or acceptability of MBCT as an intervention, have thus far excluded an important aspect of the course involving the experience of meditative homework assignments. Therefore, the aim of this study was to explore subjective accounts of the meaning of carrying out meditative homework assignments in the context of a National Health Service (NHS) run MBCT course. The research questions focused on the impact of meditative homework on thought processes as well as an exploration of barriers and facilitating factors from a participant's perspective.Six individual in-depth interviews were conducted with participants all of whom had completed the full MBCT programme. Interpretive phenomenological Analysis (IPA) was used as the methodology for analysing interview transcripts. Data analysis began with a detailed examination of one case until a thorough analysis was completed after which subsequent cases were analysed. Finally a cross case analysis was carried out where individual themes were interrogated for similarities and differences (Smith, et al., 2009).

Two master themes were presented: 'The relationship of meditative homework to metacognitive experience' and 'Motivating and discouraging factors for engagement in meditative practice'. Results reveal a transformation in metacognitive processes as a result of undertaking meditative homework. The subjective experience of metacognitive processes is examined in the context of existing psychological theories including the ICS (Teasdale, 1999a, 1999b) as well as the S-REF (Wells, 2000) theory involving metacognitions. A model for perceived facilitating factors and difficulties experienced in carrying out meditative homework is constructed based on the Integrated Theoretical Foundations Model for CBT homework assignment (Kazantzis, et al., 2005). The model explores participants' motivation in three stages of the homework process: firstly during assignment of the meditative homework task, secondly in completing the planned task and finally carrying out review of the task in question. Implications of the present study are discussed in relation to psychological literature, homework assignment and the practise of MBCT.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be 18 to 65 years of age and recruited through an NHS Trust offering MBCT.
* At present I am uncertain of the exact inclusion and exclusion criteria as the relevant NHS trust is yet to be determined, so the guidelines recommended by Teasdale et al., (2000) and Ma and Teasdale (2004) will be used.
* These authors suggest that MBCT has no significant effect on reducing the relapse rates of depression in patients with ≤ 2 episodes of depression.
* Therefore the present study will use participants who have experienced more than three episodes of depression as judged by the relevant NHS Trust.
* No restrictions are placed in terms of participants' use of antidepressant medication.

Exclusion Criteria:

* Exclusion criteria consists of disorders where the participant would have difficulties understanding and/or applying mindfulness techniques, including current alcohol or substance dependence, borderline personality disorder, organic mental disorder or pervasive developmental delay, schizoaffective disorder, schizophrenia, schizophreniform disorder, delusional disorder and psychotic disorder not otherwise specified.
* Potential participants engaging in yoga or Buddhist meditation more than twice a week are excluded as these practices significantly overlap with the MBCT program.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eight participants will be recruited from South London and Maudsley NHS Trust, which is a national health service site offering Mindfulness Based Cognitive Therapy (MBCT).
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2009-12; Primary Completion 2010-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
The project involves one 60-minute interview per participant aiming to evaluate lived experience of having taken part in an MBCT programme. The specific focus is on MBCT programme's possible impact on personal identity, barriers and facilitating factors. | Interviews are conducted upon completion of MBCT course

CONTACTS AND LOCATIONS:
Overall Officials: Marika Lahtinen, Principal Investigator — University of East London
Locations (1):
- South London & Maudsley NHS Trust, London, London, United Kingdom

REFERENCES:
- See also: Resources for Mindfulness Based Cognitive Therapy (MBCT) — http://mbct.co.uk/